CLINICAL TRIAL: NCT02508571
Title: The Effects of Direct Swallowing Training and Oral Sensorimotor Stimulation in Preterm Infants
Brief Title: Direct Swallowing Training and Oral Sensorimotor Stimulation in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ee-Kyung Kim, Clinical associate professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 1401139552
Record Dates: First submitted 2015-07-23; First posted 2015-07-27 (Estimated); Results first posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Premature Birth of Newborn; Intervention Studies
Keywords: Infant, Premature; Intervention Studies; Bottle feeding
MeSH Terms: conditions — Premature Birth; Bottle Feeding

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Allocation is concealed from all investigators, nurses, doctors, and parents, with the sole exception of the occupational therapists, who provided the interventions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Sham Comparator): Two 15-minute sessions of sham intervention/day, five days a week
  Interventions: Other: Sham intervention
- DST group (Experimental): One session of DST and the other of sham intervention/day, five days a week
  Interventions: Other: Direct swallowing training (DST); Other: Sham intervention
- DST+OSMS group (Experimental): One session of DST and the other of OSMS/day, five days a week
  Interventions: Other: Direct swallowing training (DST); Other: Oral sensorimotor stimulation (OSMS)

INTERVENTIONS:
Other: Direct swallowing training (DST) — The DST consists of placing a bolus of 0.05-0.2 mL of formula milk (if the parents refuse, distilled water) via a 1-mL syringe directly on the medial-posterior part of the tongue approximately at the level of the hard and soft palate junction. The volume is started with 0.05 mL, and increased in increments of 0.05 mL to a maximum of 0.2 mL until the swallowing reflex is observed. Once the minimal volume necessary to initiate the swallow reflex is identified, it is used for the duration of the training. The bolus is provided every 30 sec over the 15-minute program or as tolerated. It is continued until infants are able to complete independent oral feeding, 2 days in a row with no adverse events that do not self-resolve.
  Arms: DST group; DST+OSMS group
Other: Oral sensorimotor stimulation (OSMS) — The OSMS consists of a 15-minute stimulation program, whereby the first 12 minutes involve stroking the cheeks, lips, gums, and tongue, and the final 3 minutes consist of sucking on a pacifier. It is continued until infants are able to complete independent oral feeding, 2 days in a row with no adverse events that do not self-resolve.
  Arms: DST+OSMS group
Other: Sham intervention — The sham intervention consisted of the therapists placing his/her hands into the incubator or bassinet for 15 minutes without touching the infants. It is continued until infants are able to complete independent oral feeding, 2 days in a row with no adverse events that do not self-resolve.
  Arms: Control; DST group

SUMMARY:
This is randomized controlled trial investigating the effects of direct swallowing training and oral sensorimotor stimulation in preterm infants on oral feeding performance.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants : before 32+0 weeks gestation
* Infants who are receiving full tube feeding (more than 120 ml/kg/day)
* Infants who discontinue of nasal continuous positive airway pressure before postmenstrual age 33+0 weeks
* 'Feeders and growers'
* The parents of the subject voluntarily sign the informed consent

Exclusion Criteria:

* Major congenital anomalies : face, central nervous system, gastrointestine, heart, etc
* Gastrointestinal complications
* Chronic medical complications : Intraventricular hemorrhage ≥ Grade III, periventricular leukomalacia, surgical necrotizing enterocolitis

Ages: 22 Weeks to 31 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 189 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2020-09 (Actual); Study Completion 2024-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ee-kyung Kim, Principal Investigator — Seoun National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Background] Lau C, Smith EO. Interventions to improve the oral feeding performance of preterm infants. Acta Paediatr. 2012 Jul;101(7):e269-74. doi: 10.1111/j.1651-2227.2012.02662.x. Epub 2012 Apr 5. PMID 22404221
- [Background] Fucile S, Gisel E, Lau C. Oral stimulation accelerates the transition from tube to oral feeding in preterm infants. J Pediatr. 2002 Aug;141(2):230-6. doi: 10.1067/mpd.2002.125731. PMID 12183719
- [Result] Heo JS, Kim EK, Kim SY, Song IG, Yoon YM, Cho H, Lee ES, Shin SH, Oh BM, Shin HI, Kim HS. Direct swallowing training and oral sensorimotor stimulation in preterm infants: a randomised controlled trial. Arch Dis Child Fetal Neonatal Ed. 2022 Mar;107(2):166-173. doi: 10.1136/archdischild-2021-321945. Epub 2021 Jul 19. PMID 34281934

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the neonatal intensive care unit of Seoul National University Children's Hospital between July 2015 and July 2020. Infants were enrolled if they were (1) born before 32 weeks' gestation; (2) receiving full tube feeding (≥120 mL/kg/day); (3) weaned from nasal continuous positive airway pressure (NCPAP) before 33 weeks' postmenstrual age (PMA); and (4) 'feeders and growers'.
Period: Overall Study
Arm/Group | Control | DST Group | DST+OSMS Group
Started | 64 (before the start of oral feeding, 48 hours after NCPAP discontinuation) | 64 (before the start of oral feeding, 48 hours after NCPAP discontinuation) | 61 (before the start of oral feeding, 48 hours after NCPAP discontinuation)
Completed | 63 (achieved 100% oral feeds of daily intake without adverse events that did not self-resolve) | 63 (achieved 100% oral feeds of daily intake without adverse events that did not self-resolve) | 60 (achieved 100% oral feeds of daily intake without adverse events that did not self-resolve)
Not Completed | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | DST Group | DST+OSMS Group | Total
Number analyzed (Participants) | 64 | 64 | 61 | 189
Age, Continuous [Mean (Standard Deviation); unit: weeks] | 28 (1) | 29 (1) | 29 (2) | 29 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 30 | 28 | 89
  Male | 33 | 34 | 33 | 100
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  South Korea | 64 | 64 | 61 | 189

OUTCOME MEASURES:

1. Primary Outcome: Days From Start to Independent Oral Feeding
Description: Days from start to independent oral feeding (independent oral feeding, 2 days in a row with no adverse events that do not self-resolve - The first successful day)
Time Frame: From date of starting oral feeding until the date of independent, full oral feeding, an expected average of 3 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Control | DST Group | DST+OSMS Group
Number analyzed (Participants) | 63 | 63 | 60
days | 21.1 (15.3) | 17.2 (9.9) | 14.8 (9.4)

2. Secondary Outcome: Days From Start to First Full Oral Feeding
Description: first full oral feeding : The first day that attain the full oral feeding regardless of feeding side effects
Time Frame: From date of starting oral feeding until the date of first full oral feeding, an expected average of 2 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Days From Start to Complete Full Oral Feeding
Description: complete full oral feeding : 2 days in a row without any adverse events The first successful day)
Time Frame: From date of starting oral feeding until the date of complete oral full feeding, an expected average of 3-4weeks
Reporting Status: Not Posted

4. Secondary Outcome: Overall Transfer
Description: % volume taken/volume prescribed
Time Frame: Total number of assessment : 3 times ( 1. starting oral feeding, 2. volume of oral feeding/total feeding volume x 100 = 50%, 3. volume of oral feeding/total feeding volume) x 100 = 100%
Reporting Status: Not Posted

5. Secondary Outcome: Proficiency
Description: % volume taken at 5 min/volume prescribed
Time Frame: as for outcome 4
Reporting Status: Not Posted

6. Secondary Outcome: Rate of Transfer
Description: mL/min volume of milk consumed relative to the duration of the oral Feeding session
Time Frame: as for outcome 4
Reporting Status: Not Posted

7. Secondary Outcome: Volume Loss
Description: % volume of milk spilled from the lips as a percentage of the total milk transferred
Time Frame: as for outcome 4
Reporting Status: Not Posted

8. Secondary Outcome: Neonatal Oral Motor Assessment Scale (NOMAS)
Description: * comprehensive description of the infant's feeding patterns
  * identify normal oral-motor patterns and to differentiate disorganized from dysfunctional patterns
Time Frame: Total number of assessment : 2 times ( 1. 3-5 days after starting oral feeding, 2. within 3 days after stopping intervention)
Reporting Status: Not Posted

9. Secondary Outcome: Length of Hospital Stay
Description: Length of hospital stay
Time Frame: From date of admission until the date of discharge, through study completion, expected average days of 3 month
Reporting Status: Not Posted

10. Secondary Outcome: Bayley Scales of Infant and Toddler Development, Third Edition
Description: * an individually administered instrument designed to assess the developmental functioning of infants, toddlers, and young children.
  * cognitive scale, motor scale (gross motor, fine motor), language scale (receptive communication, expressive communication)
  * subtest total raw scores & scaled scores / composite scores /percentile ranks/ confidence intervals
  * Total raw score range (min~max) : cognitive (0~91), receptive communication (0~49), expressive communication (0~48), fine motor (0~66), gross motor (0~72)
  * Higher scores mean better outcomes
Time Frame: Corrected age 18-24 months
Reporting Status: Not Posted

11. Secondary Outcome: Korean Version of MacArthur-Bates Communicative Development Inventories (K M-B CDI)
Description: -a simple screening test for language development
Time Frame: postnatal age 36±2 months
Reporting Status: Not Posted

12. Secondary Outcome: Korean-Wechsler Preschool and Primary Scale of Intelligence (K-WPPSI)-Fourth Edition.
Description: * An innovative measure of cognitive development and an intelligence test for preschoolers and young children
  * Primary index scales> verbal comprehension, visual spatial, fluid reasoning, working memory, processing speed ==> Full scale IQ
  * Ancillary index scales > vocabulary acquisition
  * scaled score, composite score, percentile rank, CI
  * Range of Full scale IQ : min (40) ~ max (160)
  * Higher scores mean better outcomes.
Time Frame: aged 4:00~4:11 years
Reporting Status: Not Posted

13. Secondary Outcome: Korean Developmental Screening Test
Description: * A fill-up questionnaire to be answered by parents so as to determine who experience developmental problems
  * Domains: gross motor, fine motor, language, cognition, sociality, self-care
  * Score range of each domain : min (0) ~ max (24)
  * Higher scores mean better outcomes.
Time Frame: postnatal age 48±3 months
Reporting Status: Not Posted

14. Secondary Outcome: Strengths and Difficulties Questionnaire
Description: * a brief behavioural screening questionnaire
  * 5 subscales: Emotional problems scale, Conduct problems scale, Hyperactivity scale, Peer problems scale, Prosocial scale (score range of each scale : 0-10)
  * total difficulties score : summing scores from all the scales except the prosocial scale (score range : 0-40)
  * Lower scores mean better outcomes for the all scales except the prosocial scale
Time Frame: postnatal age 48±3 months
Reporting Status: Not Posted

15. Secondary Outcome: Behavioral Pediatrics Feeding Assessment Scale (BPFAS)
Description: * A comprehensive and widely used measure of behavioral and skill-based feeding problems
  * It consists of 35 questions: 25 related to child eating, and 10 related to parent feeding behaviors.
  * Parents answer each question on a five-point Likert scale, then indicate whether they perceive that behavior to be problematic or not.
  * Child an parent frequency scores : from the Likert scales (score range : min 35 ~ max 175)
  * Child and parent problem scores : from the yes/no questions
Time Frame: postnatal age 48±3 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: during the period in which the intervention was applied, an average of 18 days
Arm/Group | Control | DST Group | DST+OSMS Group
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/64 | 1/61
Serious Adverse Events (participants affected / at risk) | 0/64 | 0/64 | 1/61
Other Adverse Events (participants affected / at risk) | 9/64 | 5/64 | 5/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control (N=64) | DST Group (N=64) | DST+OSMS Group (N=61)
Death (Gastrointestinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=64) | DST Group (N=64) | DST+OSMS Group (N=61)
Apnea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (4) | 1 (1)
Bradycardia (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4) | 3 (5)
desaturation (Respiratory, thoracic and mediastinal disorders) | 6 (13) | 4 (5) | 2 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-01): https://cdn.clinicaltrials.gov/large-docs/71/NCT02508571/Prot_SAP_000.pdf